CLINICAL TRIAL: NCT02928081
Title: Standard Versus Extended Lymphadenectomy in Pancreatoduodenectomy
Brief Title: Standard Versus Extended Lymphadenectomy in Pancreatoduodenectomy for Patients With Pancreatic Head Adenocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Collaborators: Royal Liverpool University Hospital (Other Government)
Responsible Party: Principal Investigator, Chen Hongyu, Hongyu Chen,MD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015267
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Carcinoma, Pancreatic Ductal
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended lymphadenectomy (Experimental): In addition to the standard lymphadenectomy, the nerve tissues around CHA and the SMA and nodes around the celiac trunk and SMA (No.16a2, 16b1) must be dissected. Retroperitoneal lymphatic tissue, nerves and connective tissue range from the hepatic portal down to the beginning part of the inferior mesenteric artery, the right to the right renal hilus, left to the left edge of the abdominal aorta is included.
  Interventions: Procedure: Extended lymphadenectomy
- Standard lymphadenectomy (Other): Lymph node dissection includes the superior and inferior pyloric nodes (LN5, LN6), anterior and posterior nodes along the common hepatic artery (CHA) (LN8a, 8b), nodes along the common hepatic duct, common bile duct and cystic duct (LN12b1, 12b2, 12c), posterior pancreatoduodenal nodes (LN13a, 13b), nodes along the superior mesenteric artery (SMA) (LN14a, 14b), anterior pancreatoduodenal nodes (LN17a, 17b), but excluding the nerve tissues around common hepatic artery and the superior mesenteric artery.
  Interventions: Procedure: Standard lymphadenectomy

INTERVENTIONS:
Procedure: Extended lymphadenectomy — Extended lymphadenectomy with nerve tissues around CHA and the SMA and nodes around the celiac trunk and SMA (No.16a2, 16b1)
  Arms: Extended lymphadenectomy
Procedure: Standard lymphadenectomy — Lymph node dissection includes(LN5, LN6),(LN8a, 8b),(LN12b1, 12b2, 12c),(LN13a, 13b),(LN14a, 14b),(LN17a, 17b)
  Arms: Standard lymphadenectomy

SUMMARY:
The aim of this study is to determine whether the performance of extended lymphadenectomy in association with pancreatoduodenectomy improves the long-term survival in patients with pancreatic head ductal adenocarcinoma.Half of participants will receive pancreatoduodenectomy with extended lymphadenectomy,while the other half will receive pancreatoduodenectomy with standard lymphadenectomy.

DETAILED DESCRIPTION:
Pancreatic cancer is a common malignant disease of the digestive system, and its incidence has been steadily increasing recently. Currently, the only potential curative treatment for pancreatic cancer is radical surgery. However, due to the peculiarity of the anatomical location of pancreas (in the retroperitoneum, surrounded by peripheral nerves and blood vessels) and its biological characteristics (neurotropic, highly malignant, and with probable skip metastasis), it is difficult to achieve R0 resection in patients with pancreatic cancer. High postoperative recurrence and distant metastasis rate are key factors in reducing long-term survival of patients with pancreatic cancer. The radical surgery modalities for pancreatoduodenectomy to achieve R0 resection involve extended lymphadenectomy, multivisceral resections, with or without simultaneous vein removals. Currently, the lymphadenectomy extent and approaches used to achieve R0 status are diverse. In 2014, the International Study Group for Pancreatic Surgery (ISGPS) reached a consensus to strive to resect lymph nodes (LNs) 5, 6, 8a, 12b1, 12b2, 12c, 13a, 13b, 14a, 14b, 17a, and 17b in standard lymphadenectomy for pancreatoduodenectomy. However, no consensus was reached on dissection of LN 16 due to variation in the literature and different expert opinions. On the current evidence, benefit of extended lymph node dissection seems to be outweighed by the risks. But deficiencies exist in the design of previous RCTs, such as insufficient sample size, lack of certain critical data for statistical analysis, inclusion of other pathological types of pancreatic neoplasms and variable retroperitoneal lymph node resection and nerve plexus dissection . Therefore, the power of evidence was low. Most studies report a high frequency of lymph node metastasis to LNs 13, 14, 17, 12 and 16 in pancreatic cancer, and tendency to metastasis from LNs 13, 14 to LN 16. In a lot of case reports, only nodal station 16a2 and 16b1 were positive in LN 16.

This study is performed to confirm whether pancreatoduodenectomy with extended lymphadenectomy could improve survival. Subjects undergoing surgery will be randomized to pancreatoduodenectomy with extended lymphadenectomy including nerve tissues around CHA and the SMA and nodes around the celiac trunk and SMA (No.16a2, 16b1) versus standard pancreatoduodenectomy. Subjects will be followed every three months for survivorship or death. The primary endpoint of 5-year overall or disease-free survival survival will be determined at five year post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject was diagnosed with pancreatic ductal adenocarcinoma supported by pathological and radiological examination preoperatively
* Subject with absence of vascular invasion and metastasis
* Subject with absence of prior history of cancer

Exclusion Criteria:

* Subject was diagnosed that other pancreatic tumour types (neuroendocrine tumors, intraductal papillary mucinous neoplasm, serous cystadenoma, mucinous cystadenocarcinoma, solid pseudopapillary neoplasm and pancreatitis)
* Subject was found with liver, omental, mesenteric or peritoneal metastasis intraoperatively
* Subject with presence of other significant diseases (e.g., coronary heart disease)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-02 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival rate | 5 years
  The percentage of patients that are alive at a 5 year

SECONDARY OUTCOMES:
Postoperative pancreatic fistula | Within 30 days or before discharge
  ISGPS definition
Bile leakage | Within 30 days or before discharge
  ISGLS definition
Delayed gastric emptying | Within 30 days or before discharge
  ISGPS definition
Post-pancreatectomy haemorrhage | Within 30 days or before discharge
  ISGPS definition
Intra-abdominal infection | Within 30 days or before discharge
  Presence of fever, signs of peritonitis, high leukocytes count or positive peritoneal drainage fluid culture
Wound infection | Within 30 days or before discharge
  Requiring invasive treatment, for example: positive wound exudate culture and requiring continuous re-open drainage or invasive treatment
Postoperative mortality | Within 30 days or 60 days
  Death due to any cause before or at postoperative day 30 and 60
Quality of life | 1 or 3 or 5 year
  EORTC QLQ-C30, according to the scoring manual published by the EORTC Quality of Life group
5-year disease-free survival rate | 5 years
  The percentage of patients alive without recurrence at a 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Chen, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xiong J, Szatmary P, Huang W, de la Iglesia-Garcia D, Nunes QM, Xia Q, Hu W, Sutton R, Liu X, Raraty MG. Enhanced Recovery After Surgery Program in Patients Undergoing Pancreaticoduodenectomy: A PRISMA-Compliant Systematic Review and Meta-Analysis. Medicine (Baltimore). 2016 May;95(18):e3497. doi: 10.1097/MD.0000000000003497. PMID 27149448
- [Background] Xiong JJ, Tan CL, Szatmary P, Huang W, Ke NW, Hu WM, Nunes QM, Sutton R, Liu XB. Meta-analysis of pancreaticogastrostomy versus pancreaticojejunostomy after pancreaticoduodenectomy. Br J Surg. 2014 Sep;101(10):1196-208. doi: 10.1002/bjs.9553. Epub 2014 Jul 16. PMID 25042895
- [Result] Chen Y, Ke N, Tan C, Zhang H, Wang X, Mai G, Liu X. Continuous versus interrupted suture techniques of pancreaticojejunostomy after pancreaticoduodenectomy. J Surg Res. 2015 Feb;193(2):590-7. doi: 10.1016/j.jss.2014.07.066. Epub 2014 Aug 5. PMID 25175768
- [Result] Chen Y, Tan C, Mai G, Ke N, Liu X. Resection of pancreatic tumors involving the anterior surface of the superior mesenteric/portal veins axis: an alternative procedure to pancreaticoduodenectomy with vein resection. J Am Coll Surg. 2013 Oct;217(4):e21-8. doi: 10.1016/j.jamcollsurg.2013.07.383. No abstract available. PMID 24054418
- [Result] Chen Y, Wang X, Ke N, Mai G, Liu X. Inferior mesenteric vein serves as an alternative guide for transection of the pancreatic body during pancreaticoduodenectomy with concomitant vascular resection: a comparative study evaluating perioperative outcomes. Eur J Med Res. 2014 Aug 21;19(1):42. doi: 10.1186/s40001-014-0042-z. PMID 25141915
- [Result] Nimura Y, Nagino M, Takao S, Takada T, Miyazaki K, Kawarada Y, Miyagawa S, Yamaguchi A, Ishiyama S, Takeda Y, Sakoda K, Kinoshita T, Yasui K, Shimada H, Katoh H. Standard versus extended lymphadenectomy in radical pancreatoduodenectomy for ductal adenocarcinoma of the head of the pancreas: long-term results of a Japanese multicenter randomized controlled trial. J Hepatobiliary Pancreat Sci. 2012 May;19(3):230-41. doi: 10.1007/s00534-011-0466-6. PMID 22038501
- [Result] Jang JY, Kang MJ, Heo JS, Choi SH, Choi DW, Park SJ, Han SS, Yoon DS, Yu HC, Kang KJ, Kim SG, Kim SW. A prospective randomized controlled study comparing outcomes of standard resection and extended resection, including dissection of the nerve plexus and various lymph nodes, in patients with pancreatic head cancer. Ann Surg. 2014 Apr;259(4):656-64. doi: 10.1097/SLA.0000000000000384. PMID 24368638
- [Derived] Wang Z, Ke N, Wang X, Wang X, Chen Y, Chen H, Liu J, He D, Tian B, Li A, Hu W, Li K, Liu X. Optimal extent of lymphadenectomy for radical surgery of pancreatic head adenocarcinoma: 2-year survival rate results of single-center, prospective, randomized controlled study. Medicine (Baltimore). 2021 Sep 3;100(35):e26918. doi: 10.1097/MD.0000000000026918. PMID 34477122